CLINICAL TRIAL: NCT04436068
Title: Evaluation of Hyperfine Low Field Strength Portable Point-of-Care Magnetic Resonance Imaging System in Hydrocephalus and Other Conditions Prompting Outpatient Brain Imaging
Brief Title: Hyperfine Portable MRI in Hydrocephalus and Other Conditions Prompting Outpatient Brain Imaging
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Joel M. Stein, MD, PhD, Assistant Professor of Radiology, University of Pennsylvania
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 832913
Record Dates: First submitted 2020-06-10; First posted 2020-06-17 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Hydrocephalus; Neurological Disorder
Keywords: MRI; Magnetic Resonance Imaging; CT; Shunt
MeSH Terms: conditions — Hydrocephalus; Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Outpatients with known or suspected hydrocephalus (Experimental)
  Interventions: Device: Hyperfine MRI scan
- Outpatients with other known or suspected neurological condition (Experimental)
  Interventions: Device: Hyperfine MRI scan

INTERVENTIONS:
Device: Hyperfine MRI scan — Participants receive a Hyperfine low field strength brain MRI scan in addition to a regularly scheduled standard clinical CT or MRI scan.

SUMMARY:
Participants with known or suspected hydrocephalus will receive brain scans using the Hyperfine, low field strength, portable, magnetic resonance imaging (MRI) system in addition to their scheduled outpatient standard of care clinical computed tomography (CT) or MRI scan. The purpose of this pilot study is to evaluate the feasibility and acceptability of using the Hyperfine system in an outpatient setting and to compare its diagnostic performance to standard clinical imaging.

Outpatients with other known or suspected neurological disorders or conditions prompting routine clinical brain imaging with MRI or CT will also be enrolled and the diagnostic performance of low field scans compared to that of the same day standard of care clinical imaging.

DETAILED DESCRIPTION:
Hydrocephalus is a medical condition in which an abnormal buildup of cerebrospinal fluid (CSF) causes the fluid-filled spaces of the brain, the ventricles, to become enlarged. Enlarged ventricles and increased intracranial pressure can cause headaches, dizziness, blurred vision, cognitive impairment, gait disturbances and in severe cases even brain herniation or death. A tube or shunt can be inserted into the ventricles to drain the CSF either outside the body temporarily or into the abdominal cavity for long-term treatment. Sometimes such shunts need to be adjusted or replaced if fluid re-accumulates. Medical imaging scans, either computer tomography (CT) or magnetic resonance imaging (MRI), are used to diagnose hydrocephalus in adults and children.

The purpose of this pilot study is to assess the performance of a newly developed, portable, low-cost MRI machine (Hyperfine MRI) in diagnosing and following patients with hydrocephalus in comparison to routine clinical CT or MRI. Outpatients with known or suspected hydrocephalus with or without ventricular shunts will be recruited to undergo Hyperfine MRI in conjunction with their routine clinical imaging. We will evaluate both the feasibility and acceptability of using the Hyperfine unit in the outpatient setting as well as the performance of Hyperfine MRI images in identifying hydrocephalus and other key brain imaging features relative to routine CT and MRI.

Outpatients with other known or suspected neurological disorders or conditions prompting routine clinical brain imaging with MRI or CT will also be enrolled and the diagnostic performance of low field scans compared to that of the same day standard of care clinical imaging.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Suspected or confirmed diagnosis of hydrocephalus from Penn referring physician
* Other suspected or confirmed neurological disorder from Penn referring physician
* Routine clinical CT or MRI of the brain scheduled/obtained on the same day as Hyperfine imaging.
* Informed consent obtained from patient or legally authorized representative

Exclusion Criteria:

* Contraindications to routine 1.5T MRI evaluation, including electrical implants such as cardiac pacemakers or perfusion pumps, ferromagnetic implants such as aneurysm clips, surgical clips, protheses, artificial hearts or heart valves with steel parts, metal fragments, shrapnel, tattoos near the eye, steel implants, or other irremovable ferromagnetic objects
* History of uncontrolled seizures
* Claustrophobia
* Weight greater than or equal to 400lbs (181.4kg)
* Pregnancy
* Inability or suspected inability to comply with the study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-06-28 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Presence of hydrocephalus | Through study completion, an average of 60 minutes
  Presence or absence of hydrocephalus will be determined qualitatively based on neuroradiologist interpretation of low-field MRI scans and companion standard clinical MRI or CT scans to evaluate performance using the low-field device to make this determination.
Quantitative ventricular volumes | Through study completion, an average of 60 minutes
  Quantitative ventricular volumes (mL) will be obtained and compared for low-field and companion standard clinical MRI scans.
Presence of other important imaging findings | Through study completion, an average of 60 minutes
  Presence of other important imaging findings will be determined qualitatively based on neuroradiologist interpretation of low-field MRI scans and companion standard clinical MRI or CT scans.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No